CLINICAL TRIAL: NCT04839237
Title: The Effect and the Pharmacogenomics Study of Liraglutide in Obese Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor decides withdrawn this study.
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201710832
Record Dates: First submitted 2018-03-27; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Liraglutide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liraglutide (Experimental): Obese patients with HbA1C lower than 9.0%,receive Liraglutide alone for 3 months.
  Interventions: Drug: Liraglutide
- Liraglutide combined with metformin (Experimental): Obese patients with HbA1C ≥9.0%, receive Liraglutide in combination with metformin for 3 months.
  Interventions: Drug: Liraglutide;metformin

INTERVENTIONS:
Drug: Liraglutide — The treatment of Liraglutide lasted three months,During the first week: 0.6mg per day, subcutaneous injection;During the second week: 1.2mg per day, subcutaneous injection; From third week onwards,1.8mg per day, subcutaneous injection.
  Other Names: Victoza
  Arms: Liraglutide
Drug: Liraglutide;metformin — The treatment of Liraglutide combined with metformin lasted three months.For Liraglutide,during the first week: 0.6mg per day, subcutaneous injection;during the second week: 1.2mg per day, subcutaneous injection; from third week onwards,1.8mg per day, subcutaneous injection.For metformin,during three months:0.5g each time, 3 times per day,oral.
  Other Names: Victoza;Glucophage
  Arms: Liraglutide combined with metformin

SUMMARY:
This studay evaluates the effect of liraglutide in the treatment of obese patients ande the influence of genetic factors on the curative effect.Half of participants will receive Liraglutide alone,while the other half who can not achieving adequate glycaemic control will receive Liraglutide and metformin in combination.

DETAILED DESCRIPTION:
Background:The rapid growth of obese or overweight people in the world has become a major social problem. Obese often associated with kinds of metabolic disorders, especially type 2 diabetes, and Liraglutide can effectively reduce weight and improve blood glucose.Previous studies have indicated that most patients will experience different degrees of weight loss after using Liraglutide, but there is also a small number of patients with no significant weight loss.The gene polymorphism among individuals may affect the weight loss effect of Liraglutide.

Objectives：1.To find the relationships between genetic variants and the response of Liraglutide to treatment of obese patients.2.To investigate the effects of Liraglutide on weight, metabolism (blood glucose, blood lipid, uric acid, etc.) and gut microbiota in obese Chinese patients.

Intervention:Half of participants will receive Liraglutide alone,while the other half who can not achieving adequate glycaemic control will receive Liraglutide and metformin in combination.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 65 years (to the date of screening)；
2. The newly diagnosed obese patients (BMI greater than 28 kg/m2) or abdominal obesity (male waist circumference is greater than 90cm, female waist is greater than 85cm).
3. Nearly a month have not used weight-related drugs,including various weight-loss drugs,GLP-1 analogs or agonists,metformin, acarbose,insulin,anti hyperthyroid drugs,etc;Or recently used weight-related drugs but the stable dose was more than 1 month,and the drug dose remained constant or decreased during the trial.
4. Weight stable for more than 3 months (weight fluctuations <5%).

Exclusion Criteria:

1. Pregnant female.
2. Secondary diseases caused by other diseases: including hypothyroidism, increased cortisol, hypothalamic and pituitary lesions caused by obesity, all kinds of drug-induced obesity, and others.
3. Severe cardiovascular and cerebrovascular diseases (heart failure, myocardial infarction, acute hemorrhagic or ischemic encephalopathy), pulmonary heart disease or pulmonary insufficiency, renal failure, severe hepatitis.
4. Combined with acute complications of diabetes such as ketoacidosis, lactic acidosis, hyperosmolar state of diabetes.
5. Nearly a month had surgery, trauma, infection and so on.
6. Limb deformity incomplete, difficult to accurately determine the height, weight and other physical indicators.
7. Poor medication compliance or serious side effects (severe rash, syncope, etc.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Weight Change at 3 months | baseline and 3 months
  Measured in kilograms
Genotype | baseline

SECONDARY OUTCOMES:
Change in waist circumference | baseline and 3 months
  Measured in cm
Change in systolic blood pressure | baseline and 3 months
  Measured in mmHg
Change in diastolic blood pressure | baseline and 3 months
  Measured in mmHg
Change in HbA1c | baseline and 3 months
  Measured in %
Change in plasma glucose | baseline and 3 months
  Measured in mmol/l
Change in insulin | baseline and 3 months
  Measured in μU/ml
Change in lipids-total cholesterol | baseline and 3 months
  Measured in mmol/l
Change in lipids-low density lipoprotein cholesterol | baseline and 3 months
  Measured in mmol/l
Change in lipids-high density lipoprotein cholesterol | baseline and 3 months
  Measured in mmol/l
Change in lipids-triglycerides | baseline and 3 months
  Measured in mmol/l
Change in lipids-free fatty acids | baseline and 3 months
  Measured in μmol/l
Change in Uric Acid | baseline and 3 months
  Measured in mmol/l
Gut microbiota composition | 3 months
  Gut microbiota composition is assessed by 16S rRNA pyrosequencing. This analysis allows to obtain the relative abundance (%) of the different bacterial taxa and OTUs (operational taxonomic units).

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China